CLINICAL TRIAL: NCT02147184
Title: Serotonin Reuptake Inhibitors and Bone Mineralization in Adolescents
Brief Title: Do Serotonin Reuptake Inhibitors (SSRIs) Affect Bone Mass in Adolescents
Acronym: SSRI_BMD
Status: Completed | Type: Observational
Sponsor: Chadi A. Calarge (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Chadi A. Calarge, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201109866; R01MH090072-01A1 (NIH)
Record Dates: First submitted 2014-04-02; First posted 2014-05-26 (Estimated); Results first posted 2017-10-24 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: The Skeletal Effects of SSRIs
Keywords: SSRI; serotonin transporter; DXA; pQCT; bone mass; adolescents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum plasma DNA whole blood Stools Urine Paxgene
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SSRI Group: Participants within one month of starting an SSRI
- Unmedicated Group: No treatment with SSRIs

SUMMARY:
Building on findings from animal studies, pediatric clinical trials, epidemiologic research in adults, and on preliminary findings from the investigators' laboratory in children and adolescents, this project aims to investigate whether selective serotonin reuptake inhibitors (SSRIs), a group of widely-used psychotropics, are associated with impaired bone mineralization in youths. Establishing such an association is a first step in a process that would eventually involve developing preventative interventions. Identifying genetic factors that place certain youths at higher risks for this side effect would ultimately allow clinicians to tailor treatment to the needs and vulnerabilities of each youth, moving the field closer towards individualized medicine.

DETAILED DESCRIPTION:
Bone mass achieved by early adulthood is a major determinant of lifetime risk for osteoporosis. Therefore, optimizing peak bone mass is crucial to avoiding bone fracture with its associated morbidity and mortality.

Emerging evidence suggests that serotonin plays a central role in bone metabolism. For example, preclinical experiments have shown that bone cells express the serotonin transporter and a variety of functional serotonin receptors whose activity modulates bone turnover. Epidemiologic studies have linked SSRIs to reduced bone mineral density and increased fracture risk in the elderly. SSRIs are widely used in youths to treat a number of psychiatric disorders. However, while their short-term efficacy and safety have been established, their long-term safety remains little investigated.

The investigators aim to recruit, in a 2-year prospective observational study, 15 to 20 year-old participants upon the initiation of SSRI treatment. During the study period, bone mineral density of the lumbar spine and whole body will be measured using dual-energy x-ray absorptiometry (DXA) and of the radius using peripheral quantitative computed tomography (pQCT). A detailed psychiatric assessment will be conducted to control for psychopathology, as a potential confounding factor affecting bone mineralization. Changes in psychiatric treatment during the follow up period will also be documented and accounted for. By using a group of controls, of comparable age and sex distribution, the investigators aim to evaluate 1) whether psychopathology, at baseline, is associated with low bone mass, 2) if treatment with SSRIs suppresses bone mineralization, and 3) if the discontinuation of the SSRI is followed by a restoration of bone mineral accrual. 4) Furthermore, genetic testing will investigate whether variants of the serotonin system genes moderate the effect of SSRI treatment on bone mineral density.

In sum, this work aims to improve the long-term safety of psychiatric treatments in order to optimize functioning and the quality of life of those who suffer from psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15 to 20 years old (inclusive).
2. Treatment with an SSRI, regardless of the indication, having been started within one month. This criterion does not apply to controls. SSRIs include: fluoxetine, citalopram, escitalopram, sertraline, paroxetine, and fluvoxamine.
3. Ability to provide consent.

Exclusion Criteria:

1. Age- and sex-adjusted height Z-score < -2 or > 2.
2. Concomitant treatment with other antidepressants, psychostimulants, or mood stabilizers and antipsychotics. Treatment with benzodiazepines, low dose trazodone, alpha-2 agonists, and antihistaminergic agents will be allowed.
3. Presence of illicit drug and/or alcohol dependence.
4. Pregnancy.
5. Primary bone diseases (e.g., Paget's disease, osteogenesis imperfecta, rheumatoid arthritis).
6. Potential secondary bone disease (e.g., due to chronic inflammatory diseases, diabetes, hypo- or hyperparathyroidism, hyperthyroidism, growth hormone deficiency, and other endocrine disturbances, history of childhood cancer, or prior transplantation).
7. Chronic disorders involving a vital organ (heart, lung, liver, kidney, brain) and congenital disorders.
8. Malnutrition conditions (e.g., chronic diarrhea, inflammatory bowel disease) or lead poisoning.
9. Chronic use of drugs affecting bone metabolism (e.g., oral corticosteroids).
10. Inability to cooperate with the BMD measurements.
11. Eating disorders, due to their potential effect on BMD.
12. If a senior in high school, plan to join an out-of-state college.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients within one month of initiating treatment with SSRIs will be recruited, regardless of the indication for SSRIs.
  Unmedicated controls will be also recruited.
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadi Calarge, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Ezenwabachili I, Deumic Shultz E, Mills JA, Ellingrod V, Calarge CA. Examining Whether Genetic Variants Moderate the Skeletal Effects of Selective Serotonin Reuptake Inhibitors in Older Adolescents and Young Adults. J Child Adolesc Psychopharmacol. 2023 Sep;33(7):260-268. doi: 10.1089/cap.2023.0007. Epub 2023 Aug 9. PMID 37579130
- [Derived] Martins LB, Delevati Colpo G, Calarge CA, Teixeira AL. Inflammatory Markers Profile in Older Adolescents During Treatment with Selective Serotonin Reuptake Inhibitors. J Child Adolesc Psychopharmacol. 2021 Aug;31(6):439-444. doi: 10.1089/cap.2020.0140. Epub 2021 Jun 24. PMID 34166063
- [Derived] Mellick WH, Mills JA, Kroska EB, Calarge CA, Sharp C, Dindo LN. Experiential Avoidance Predicts Persistence of Major Depressive Disorder and Generalized Anxiety Disorder in Late Adolescence. J Clin Psychiatry. 2019 Oct 22;80(6):18m12265. doi: 10.4088/JCP.18m12265. PMID 31644841
- [Derived] Dindo LN, Recober A, Haddad R, Calarge CA. Comorbidity of Migraine, Major Depressive Disorder, and Generalized Anxiety Disorder in Adolescents and Young Adults. Int J Behav Med. 2017 Aug;24(4):528-534. doi: 10.1007/s12529-016-9620-5. PMID 28032323
- [Derived] Deumic E, Butcher BD, Clayton AD, Dindo LN, Burns TL, Calarge CA. Sexual Functioning in Adolescents With Major Depressive Disorder. J Clin Psychiatry. 2016 Jul;77(7):957-62. doi: 10.4088/JCP.15m09840. PMID 27464316

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 09/2010 and 12/2014, 287 participants were recruited into this longitudinal observational study, from outpatient and inpatient clinical settings as well as by advertisement and word of mouth.
  However, 23 of them either did not complete their intake visit or had to be excluded due to discovery of exclusionary conditions.
Pre-assignment Details: within one month of starting a SSRI or taking no psychotropics
Period: Overall Study
Arm/Group | SSRI Group | Unmedicated Group
Started | 127 | 137
Completed | 78 | 110
Not Completed | 49 | 27
Not completed — Lost to Follow-up | 28 | 15
Not completed — Study Burden | 11 | 7
Not completed — Pregnancy | 6 | 0
Not completed — Moved out of state | 3 | 3
Not completed — Physician Decision | 0 | 2
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SSRI Group | Unmedicated Group | Total
Number analyzed (Participants) | 127 | 137 | 264
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.8 (1.7) | 19.0 (1.5) | 18.9 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 76 | 159
  Male | 44 | 61 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 22
  Not Hispanic or Latino | 116 | 126 | 242
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 4 | 11 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 114 | 119 | 233
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 127 | 137 | 264

OUTCOME MEASURES:

1. Primary Outcome: Total Body Less Head Bone Mineral Content (TBLH BMC) Z-score (Adjusted for Age-sex-height-race)
Description: Whole-body dual energy x-ray absorptiometry (DXA) scan was obtained using a Hologic QDR DELPHI-4500A unit or a Hologic Discovery A unit (Hologic, Inc, Bedford, MA). The two DXA units were cross-calibrated.
Time Frame: At baseline and every 8 months up to 2 years.
Population: These are the starting sample size but the figures below reflect participant attrition.
Measure: Mean (Standard Deviation); unit: Z score (age-sex-height-race specific)
Arm/Group | SSRI Group | Unmedicated Group
Number analyzed (Participants) | 127 | 137
Z score (age-sex-height-race specific)
  Baseline | 0.35 (0.84) | 0.43 (0.90)
  8 Months: number analyzed (Participants) | 75 | 106
  8 Months | 0.36 (0.84) | 0.44 (0.92)
  16 Months: number analyzed (Participants) | 63 | 87
  16 Months | 0.32 (0.87) | 0.47 (0.90)
  24 Months: number analyzed (Participants) | 76 | 108
  24 Months | 0.32 (0.90) | 0.41 (0.87)

2. Primary Outcome: Trabecular Volumetric Bone Mineral Density at the Ultradistal Radius
Description: Volumetric bone mineral density (vBMD) at the nondominant radius (4% and 20% sites) was measured, at study entry and every four months, with peripheral quantitative computed tomography (pQCT), using a Stratec XCT-2000 scanner (Stratec, Inc., Pforzheim, Germany). Image analysis was performed using the manufacturer's software package, version 6.0. pQCT scans compromised by movement were rejected. Quality control and calibration of the equipment were performed daily.
Time Frame: At baseline and every 4 months up to 2 years.
Population: This was the starting sample size. However, the figures below reflect participant attrition and exclusion of scans due to movement artifact.
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | SSRI Group | Unmedicated Group
Number analyzed (Participants) | 127 | 137
mg/cm^3
  Baseline: number analyzed (Participants) | 121 | 133
  Baseline | 213.7 (37.7) | 220.7 (35.0)
  4 Months: number analyzed (Participants) | 88 | 109
  4 Months | 212.9 (40.7) | 220.0 (37.8)
  8 Months: number analyzed (Participants) | 73 | 101
  8 Months | 217.9 (40.2) | 220.8 (39.5)
  12 Months: number analyzed (Participants) | 66 | 100
  12 Months | 213.6 (42.9) | 218.9 (38.9)
  16 Months: number analyzed (Participants) | 61 | 83
  16 Months | 216.5 (40.3) | 220.9 (41.1)
  20 Months: number analyzed (Participants) | 51 | 70
  20 Months | 213.6 (41.9) | 218.7 (39.4)
  24 Months: number analyzed (Participants) | 72 | 104
  24 Months | 209.1 (40.48) | 221.7 (37.1)

3. Primary Outcome: Osteocalcin to C-terminal Telopeptide Ratio
Description: Osteocalcin (ng/mL) is a bone formation marker and C-terminal telopeptide (ng/mL) a marker of bone resorption.
Time Frame: At baseline and every 4 months up to 2 years.
Population: The figures below may be lower based on availability of serum, performance of the assay, and premature attrition.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | SSRI Group | Unmedicated Group
Number analyzed (Participants) | 127 | 137
Ratio
  Baseline: number analyzed (Participants) | 123 | 132
  Baseline | 49.1 (16.4) | 50.4 (18.7)
  4 Months: number analyzed (Participants) | 82 | 108
  4 Months | 53.9 (33.6) | 47.2 (17.3)
  8 Months: number analyzed (Participants) | 66 | 96
  8 Months | 49.7 (17.1) | 49.1 (18.2)
  12 Months: number analyzed (Participants) | 71 | 100
  12 Months | 53.4 (22.8) | 47.2 (18.1)
  16 Months: number analyzed (Participants) | 53 | 73
  16 Months | 51.9 (17.9) | 50.3 (20.9)
  20 Months: number analyzed (Participants) | 49 | 70
  20 Months | 46.8 (14.2) | 50.3 (20.8)
  24 Months: number analyzed (Participants) | 67 | 85
  24 Months | 54.5 (21.7) | 48.0 (16.5)

4. Primary Outcome: Bone-specific Alkaline Phosphatase to C-terminal Telopeptide Ratio
Description: Bone-specific alkaline phosphatase (ng/mL) is a marker of bone formation while C-terminal telopeptide (ng/mL) is a marker of bone resorption.
Time Frame: At baseline and every 4 months up to 2 years.
Population: The figures below might be less than the stated numbers above depending on availability of serum samples, the performance of the assay, and premature attrition.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | SSRI Group | Unmedicated Group
Number analyzed (Participants) | 127 | 137
Ratio
  Baseline: number analyzed (Participants) | 120 | 125
  Baseline | 49.4 (16.4) | 50.3 (18.6)
  4 Months: number analyzed (Participants) | 77 | 99
  4 Months | 54.8 (34.4) | 46.5 (16.3)
  8 Months: number analyzed (Participants) | 57 | 81
  8 Months | 51.9 (16.9) | 48.9 (16.1)
  12 Months: number analyzed (Participants) | 69 | 98
  12 Months | 54.2 (22.6) | 47.2 (18.1)
  16 Months: number analyzed (Participants) | 47 | 64
  16 Months | 52.7 (18.7) | 51.4 (21.1)
  20 Months: number analyzed (Participants) | 48 | 68
  20 Months | 46.8 (14.3) | 50.0 (20.9)
  24 Months: number analyzed (Participants) | 59 | 75
  24 Months | 56.0 (22.4) | 47.3 (14.9)

5. Secondary Outcome: Lumbar Spine Bone Mineral Density (BMD) Z-score
Description: This is a Z-score adjusted for sex, age, race, and height.
Time Frame: At baseline and every 8 months up to 2 years.
Population: This was the initial sample size per group but the figures below reflect attrition or data excluded due to artifact.
Measure: Mean (Standard Deviation); unit: Z-score (Age-Sex-Height-Race Specific)
Arm/Group | SSRI Group | Unmedicated Group
Number analyzed (Participants) | 127 | 137
Z-score (Age-Sex-Height-Race Specific)
  Baseline | -0.00 (1.03) | 0.09 (1.09)
  8 Months: number analyzed (Participants) | 74 | 106
  8 Months | 0.01 (1.06) | 0.13 (1.09)
  16 Months: number analyzed (Participants) | 63 | 87
  16 Months | -0.02 (1.19) | 0.11 (1.17)
  24 Months: number analyzed (Participants) | 76 | 108
  24 Months | 0.03 (1.18) | 0.09 (1.06)

6. Secondary Outcome: Cortical Volumetric BMD at 20% Radius
Time Frame: At baseline and every 4 months up to 2 years.
Population: This was the original sample size per group but the figures below reflect attrition and data exclusion due to movement artifacts.
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | SSRI Group | Unmedicated Group
Number analyzed (Participants) | 127 | 137
mg/cm^3
  Baseline: number analyzed (Participants) | 121 | 131
  Baseline | 1155.6 (33.0) | 1156.2 (34.5)
  4 Months: number analyzed (Participants) | 89 | 107
  4 Months | 1159.8 (29.9) | 1161.7 (29.5)
  8 Months: number analyzed (Participants) | 72 | 102
  8 Months | 1163.1 (26.7) | 1164.7 (28.5)
  12 Months: number analyzed (Participants) | 71 | 101
  12 Months | 1168.3 (26.5) | 1166.8 (27.1)
  16 Months: number analyzed (Participants) | 61 | 85
  16 Months | 1170.1 (22.6) | 1169.5 (24.9)
  20 Months: number analyzed (Participants) | 51 | 73
  20 Months | 1172.8 (27.2) | 1173.1 (22.7)
  24 Months: number analyzed (Participants) | 73 | 106
  24 Months | 1173.4 (23.0) | 1170.5 (25.4)

7. Secondary Outcome: Cortical Thickness at 20% Radius
Description: This is cortical thickness as measured by pQCT.
Time Frame: At baseline and every 4 months up to 2 years.
Population: The figures below may be lower than the overall numbers above due to exclusions for movement artifacts and premature drop outs.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | SSRI Group | Unmedicated Group
Number analyzed (Participants) | 127 | 137
mm
  Baseline: number analyzed (Participants) | 121 | 131
  Baseline | 2.70 (0.34) | 2.80 (0.35)
  4 Months: number analyzed (Participants) | 89 | 107
  4 Months | 2.68 (0.32) | 2.80 (0.34)
  8 Months: number analyzed (Participants) | 72 | 102
  8 Months | 2.72 (0.34) | 2.83 (0.36)
  12 Months: number analyzed (Participants) | 71 | 101
  12 Months | 2.69 (0.33) | 2.82 (0.36)
  16 Months: number analyzed (Participants) | 61 | 85
  16 Months | 2.72 (0.31) | 2.81 (0.36)
  20 Months: number analyzed (Participants) | 51 | 73
  20 Months | 2.72 (0.33) | 2.79 (0.35)
  24 Months: number analyzed (Participants) | 73 | 106
  24 Months | 2.67 (0.30) | 2.84 (0.38)

ADVERSE EVENTS:
Time Frame: 2 years.
Description: This was not a clinical intervention. Adverse events were simply related to participating in a study.
Arm/Group | SSRI Group | Unmedicated Group
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/137
Serious Adverse Events (participants affected / at risk) | 0/127 | 1/137
Other Adverse Events (participants affected / at risk) | 19/127 | 27/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSRI Group (N=127) | Unmedicated Group (N=137)
Fainting (Cardiac disorders) | 0 (0) | 1 (1) — Fainting during blood draw with convulsion. Neurology consult determined that it was a vasovagal reaction
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSRI Group (N=127) | Unmedicated Group (N=137)
Multiple blood draws required (Blood and lymphatic system disorders) | 10 (10) | 17 (17)
Lightheadedness (Cardiac disorders) | 6 (7) | 9 (9)
Syncope (Cardiac disorders) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was not randomized. It may not have been of a long enough duration. Measuring bone mass in lower extremities may have been necessary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No